CLINICAL TRIAL: NCT07208110
Title: Factors Associated With Mortality by Trauma in the Intensive Care Unit in Villavicencio, Colombia. A Trial Based on a Discharge Registry.
Brief Title: Mortality of Trauma in the Intensive Care Unit.
Acronym: MOTRAM-ICU-COL
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other); Clínica Primavera (Unknown)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, Principal investigator, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2025_01_QX_UCI_TMA
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Trauma (Including Fractures); Trauma ICU Patients; Trauma Injury; Trauma Patients in ICU; Trauma Patients
Keywords: Trauma; Wounds and Injuries; Intensive Care Units; Trauma Registry; Low-Middle Income Countries; Colombia
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma: Records of patients admitted to the ICU with a diagnosis of trauma, major trauma, polytrauma, severe trauma.
  Interventions: Other: Exposed to trauma
- Non-trauma: Records of patients admitted to the ICU with other non-trauma diagnosis.
  Interventions: Other: Not exposed

INTERVENTIONS:
Other: Exposed to trauma — Patients exposed to trauma previous to the admission to the ICU.
  Groups: Trauma
Other: Not exposed — Patients not exposed to trauma previous to the admission to the ICU.
  Groups: Non-trauma

SUMMARY:
In this study, it was planned to establish the factors associated with severe trauma discharged from the intensive care unit and mortality. A cross-sectional trial will be conducted to review the ICU discharge database at a two-year interval to review records of trauma admissions patients and compare them with other types of admissions. Participant institutions are general hospitals (public and private) from the Colombian Orinoco region. the prevalence of admission by trauma will also be determined.

DETAILED DESCRIPTION:
Introduction Trauma is the main cause of mortality and disability in young population worldwide. The violence and vehicle accidents are the most common mechanism, depending on regional context. Severe cases require admission to the intensive care unit usually. Comprehension of such the factors associated with trauma mortality will allow to optimize, prioritize and improve limited resources, by stratifying the risk, and focus therapeutic strategies, with a potential reduction on mortality, cost, and sequalae. The study aims to analyze the factors associated with outcomes in patients with severe trauma admitted to the intensive care unit.

Methodology An analytical cross-sectional trial will be performed, based on the review of discharge database in the intensive care unit during the period of study. The study will be performed in Hospital Departamental de Villavicencio and Clinica Primavera from January 2022 and December 2024. Al records from discharges will be reviewed to establish those related to trauma indications; the records will be divided in two groups for comparisons between the care after trauma and other admissions. Demographic variables of severity and diagnosis will be analyzed. The outcomes to evaluate will be mortality and ICU length of stay.

Expected results The cause of admission by trauma, severity scores by diagnostic groups, and the outcomes by type of trauma will be highlighted with this trial. With the advance of this research, we expect that predictive variables for mortality in trauma, polytrauma, and major trauma in the ICU, will be revealed, and a predictive model adjusted to the local context of the population cared will be established.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the intensive care unit.

Exclusion Criteria:

* None.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Records of patient discharged from the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Discharge by death or within 30 days of ICU length of stay.

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  Length of stay in the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez Gutierrez, MD, Study Director — Universidad Cooperativa de Colombia; Hospital Departamental de Villavicencio; Clínica Primavera
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No
The dataset contains reserved information of patients.

REFERENCES:
- [Result] Wang F, Li ZM, Ma T. Construction and validation of a nomogram prediction model for the need for intensive care unit admission after hip fracture surgery. Medicine (Baltimore). 2025 Jun 13;104(24):e42793. doi: 10.1097/MD.0000000000042793. PMID 40527820
- [Result] Valcarcel CR, Bieler D, Bass GA, Gaarder C, Hildebrand F; ESTES Polytrauma Consensus Group. ESTES recommendations for the treatment of polytrauma-a European consensus based on the German S3 guidelines for the treatment of patients with severe/multiple injuries. Eur J Trauma Emerg Surg. 2025 Apr 11;51(1):171. doi: 10.1007/s00068-025-02852-4. PMID 40214785
- [Result] Nunes Dos Santos MS, Stayt LC. The effectiveness of FOUR score versus GCS scale in predicting mortality and morbidity in traumatic brain injured patients in intensive care: A systematic review. Intensive Crit Care Nurs. 2025 Aug;89:104048. doi: 10.1016/j.iccn.2025.104048. Epub 2025 May 7. PMID 40339389
- [Result] Chen Y, Wei X, Sun X, Mo X, Tu J, Xie T. Development and validation of a practical predicting model for early mortality in polytrauma patients: secondary analysis from Switzerland. BMJ Open. 2025 Jun 12;15(6):e100417. doi: 10.1136/bmjopen-2025-100417. PMID 40506077
- [Result] Hefny AF, Idris K, Eid HO, Abu-Zidan FM. Factors affecting mortality of critical care trauma patients. Afr Health Sci. 2013 Sep;13(3):731-5. doi: 10.4314/ahs.v13i3.30. PMID 24250314
- [Result] Fukuchi M, Nakajima M, Fukai Y, Miyazaki T, Masuda N, Sohda M, Manda R, Tsukada K, Kato H, Kuwano H. Increased expression of c-Ski as a co-repressor in transforming growth factor-beta signaling correlates with progression of esophageal squamous cell carcinoma. Int J Cancer. 2004 Mar 1;108(6):818-24. doi: 10.1002/ijc.11651. PMID 14712482